CLINICAL TRIAL: NCT05722080
Title: E3CAPS: Improvement of the Safety of Care in Cataract Surgery Teaching on Eyesi Simulator: Learning Curve and Impact of Sleep Deprivation on Residents in Ophthalmology
Brief Title: Improvement of the Safety of Care in Cataract Surgery Teaching on Eyesi Simulator (E3CAPS)
Acronym: E3CAPS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nantes University Hospital (Other)
Collaborators: University Hospital, Tours (Other); Rennes University Hospital (Other); University Hospital, Angers (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: AP_JBD_001
Record Dates: First submitted 2022-12-22; First posted 2023-02-10 (Actual); Last update posted 2024-02-15 (Actual); Status verified 2024-02

CONDITIONS: Surgery-Complications; Cataract
Keywords: Ophthalmologic Surgical Procedures; Cataract; simulation training; Eyesi simulator; learning curve; sleep; deprivation; professionalism
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Intervention Model Description: First arm to model the learning curve of opthalmologist residents Second arm to show the impact of sleep deprivation on the surgical performance of experienced opthalmologist residents
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- simulator Eyesi - new residents (Other): Eyesi simulator learning curve for new ophthalmology residents
  Interventions: Other: Eyesi simulator
- simulator Eyesi/sleep deprivation -confirmed residents (Other): See how experienced residents perform after sleep deprivation using the Eyesi simulator
  Interventions: Other: Sleep deprivation

INTERVENTIONS:
Other: Eyesi simulator — Eyesi simulator learning curve for new ophthalmology residents
  Arms: simulator Eyesi - new residents
Other: Sleep deprivation — See how experienced residents perform after sleep deprivation using the Eyesi simulator
  Arms: simulator Eyesi/sleep deprivation -confirmed residents

SUMMARY:
The aim of this project is to reduce the risks of cataract surgery using the EyeSi simulator Axis 1: to model the learning curve of novice residents in Ophthalmology who follow the training program recommended by the "Collège des Ophtalmologistes niversitaires de France" (COUF) in order to help creating a "licence to operate" Axis 2: to evaluate the impact of sleep deprivation on the surgical performance of experienced residents in Ophthalmology

DETAILED DESCRIPTION:
Axis 1 (15 residents): Learning curve Each resident will perform four 2-hour learning sessions, under the supervision of an experienced cataract surgery trainer. Each resident will perform a standardized assessment at the beginning of the first session with the collection of scores at each surgical stage and the calculation of an average score simulating a complete surgery. This standardized assessment will then be repeated at the end of each of the 4 training sessions. These five points of measurement will make it possible to produce a learning curve for each surgical stage and for the average score simulating a complete surgery.

Axis 2 (25 residents): Sleep deprivation

* 1st session: In order to include the "experienced" residents and to limit the bias related to the learning curve of the cognitive tests and the surgical procedure

  * 3 normed assessments in autonomy to determine the average score for each resident
  * 3 trials of the Test for Attentional Performance (TAP) with parallel versions to limit test-retest learning bias
* 2nd session: No sleep deprivation

  * Sleep assessment by actimetry the night before the session (MotionWatch 8©, camntech®, validated as an alternative method to the reference method which is polysomnography)
  * Epworth sleepiness score
  * Visual Analogue Scale for Self-Rated Fatigue
  * Attentional performance tests TAP
  * 3 standardized evaluations on Eyesi in the morning and in the afternoon
* 3rd session: sleep deprivation (< 7 hours) after a working day

  * Sleep evaluation by actimetry the night before the session (MotionWatch 8©, camntech®)
  * Epworth sleepiness score
  * Self-rated visual analogue scale for fatigue
  * Attentional performance tests TAP
  * 3 Eyesi standardized evaluations in the morning and in the afternoon

ELIGIBILITY:
Inclusion Criteria:

* Novice resident in Ophthalmology (Axis 1)
* Experienced resident in Opthalmology (Axis 2 )

Exclusion Criteria:

* N/A

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-01-09 (Actual); Primary Completion 2025-01-09 (Estimated); Study Completion 2025-01-09 (Estimated)

PRIMARY OUTCOMES:
Scores on standardized simulator Eyesi assessments | Change the score from Baseline at 1 year
  Average score of standardized evaluations on EyeSi simulator. The scale title is "EyeSi score". The scores range from 0 to 100, better outcome being positively correlated with a higher score
Scores on standardized simulator Eyesi assessments after sleep deprivation | Change the score from Baseline at 1 year
  Average score of standardized evaluations on EyeSi simulator after sleep deprivation. The scale title is "EyeSi score". The scores range from 0 to 100, better outcome being positively correlated with a higher score

CONTACTS AND LOCATIONS:
Overall Officials: Pierre Lebranchu, M.D, Principal Investigator — Nantes University Hospital
Locations (2):
- France (2):
  - CHU Nantes, Nantes
  - CHU Tours, Tours

REFERENCES:
- [Derived] Ducloyer JB, Poinas A, Duchesne L, Caillet P, Ivan C, Lejus-Bourdeau C, Limousin N, Desmidt T, Pladys P, Pisella PJ, Bernard A, Lardy H, Gohier P, Martin L, Mouriaux F, Lebranchu P, Khanna RK; E3CAPS Group. Educational Concerns About the Safety of Cataract Surgery During Residency: The E3CAPS Pedagogic Study. Ophthalmol Ther. 2023 Oct;12(5):2801-2812. doi: 10.1007/s40123-023-00774-1. Epub 2023 Aug 2. PMID 37531031